CLINICAL TRIAL: NCT02907060
Title: Propess® Versus Double Balloon for Cervical Ripening of Prolonged Pregnancies: a Randomised Controlled Trial
Brief Title: Mechanical cervicAl ripeninG for Women With PrOlongedPregnancies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAGPOP
Record Dates: First submitted 2016-09-06; First posted 2016-09-20 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Prolonged Pregnancy
Keywords: prolonged pregnancy; mechanical cervical ripening
MeSH Terms: conditions — Pregnancy, Prolonged

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical cervical ripening (Experimental): mechanical cervical ripening with a Cook® Cervical Ripening Balloon
  Interventions: Device: Mechanical cervical ripening
- Pharmacological cervical ripening (Active Comparator): pharmacological cervical ripening with a 10mg slow releasing system of Dinoprostone (Propess®)
  Interventions: Drug: Pharmacological cervical ripening

INTERVENTIONS:
Device: Mechanical cervical ripening — The mechanical cervical ripening is a double transcervical balloon. The device used in the study is the Cook® Cervical Ripening Balloon with CE marked (commercialized by the Cook® laboratory, ref JCRBS-184000). It is a silicone double balloon catheter. Maximum balloon inflation is 80 mL/balloon.
  It will be used in accordance with user manual
  Arms: Mechanical cervical ripening
Drug: Pharmacological cervical ripening — The comparative pharmacological procedure is a vaginal slow releasing system of dinoprostone. The form used in the study is Propess (Ferring pharmaceuticals) containing 10mg of dinoprostone (prostaglandin E2).
  It will be used in accordance with Summary of Product Characteristics
  Arms: Pharmacological cervical ripening

SUMMARY:
A pregnancy is considered ''prolonged'' from 41 weeks of gestation. Prolonged Pregnancies (PP) are associated with increased maternal morbidity: emergency caesarean, 3rd and 4th degree perineal lesions and postpartum haemorrhage. Foetuses are at increased risk of oligohydramnios, meconium-staining and Fetal Heart Rate (FHR) anomalies. Around 15% of all pregnancies are prolonged.

A Cochrane review on induction of labour showed that a policy of labour induction at or beyond 41 weeks was associated with significantly fewer perinatal deaths. Thus the French College of Obstetricians and Gynaecologists stated, "induction of labour can be proposed to patients between 41+0 and 41+6 weeks of gestation". In cases where labour is induced and cervix is unfavourable, cervical ripening is advised. Methods of cervical ripening include pharmacological (prostaglandins) and mechanical (Foley catheter or trans-cervical double balloon) methods. Those two methods were compared in the PROBAAT trial among women with term pregnancies (beyond 37+0). The rates of caesarean section with these two strategies were identical, however uterine hyper stimulation with FHR anomalies occurred less when cervical ripening was mechanical.

Considering pharmacological cervical ripening is associated with more uterine hyper stimulation and more FHR anomalies, it may not be the most appropriate in cases of fragile foetuses that include cases of prolonged pregnancies. Considering prolonged pregnancies are associated with a risk of FHR anomalies and that cervical ripening with a pharmacological method is another factor which increases this risk: women with prolonged pregnancies could benefit from a more "gentle" cervical ripening.

At present, no particular method is recommended in cases of cervical ripening and prolonged pregnancies. We hypothesise that, in cases of prolonged pregnancies, mechanical cervical ripening, with less uterine hyperstimulation and fewer FHR anomalies, could be more appropriate and could reduce the rate of caesarean section for suspicion of fetal distress.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* ≥ 18 years old
* With a singleton cephalic pregnancy between ≥41+0 weeks and ≤ 42+0 weeks of gestation
* Gestational age estimated from the first trimester ultrasound (realized between 11 and 13+6 weeks of gestation)
* With a decision of induction of labour
* Written informed consent obtained from subject
* Subject covered by or having the rights to the French Social Security system

Exclusion Criteria:

* Bishop score ≥ 6 (favourable cervix)
* Non cephalic presentation (breech, transverse)
* Severe preeclampsia defined as the presence of preeclampsia with at least one of the following items :

  * Severe maternal hypertension (systolic blood pressure ≥ 160 mm Hg and/or diastolic blood pressure ≥ 110 mm Hg)
  * Renal failure with oliguria (< 500 ml/24h) or creatinine > 135μmol/L, or proteinuria > 5 g/day
  * Pulmonary oedema, epigastric pain or HELLP syndrom (hemolysis, elevated liver enzyme, low platelets)
  * Eclampsia or neurologic persisting symptoms (visual disturbances, headache, increased reflexes)
  * Thrombopenia < 100 G/L
* Prior caesarean section or uterine scar
* Placenta praevia
* Suspected genital herpes infection
* Known VIH seropositivity (confirmed by blood serology)
* Premature rupture of membranes (PROM - continual leaking of amniotic fluid or positive test in favour of PROM)
* Foetus with suspected severe congenital abnormalities
* Pathological fetal heart rate
* Contra-indications to Propess®
* Contra-indications for using Cook® Cervical Ripening Balloon
* Women under guardianship or trusteeship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1224 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Caesarean section rate for non-reassuring fetal status. | Up to 2 days after cervical ripening
  Indication of the caesarean section will be settled by an adjudication committee at the end of the study

SECONDARY OUTCOMES:
Time between cervical ripening and delivery in hours | Up to 2 days after cervical ripening
  Evaluation of time between cervical ripening and delivery in hours
Delivery rate after 12 and 24 hours of cervical ripening | up to 2 days after cervical ripening
  Evaluation of delivery rate after 12 and 24 hours of cervical ripening
Induction with oxytocin | up to 2 days after cervical ripening
  yes/no
Total dose of oxytocin required for induction of labour | up to 2 days after cervical ripening
  evaluation of total dose of oxytocin required for induction of labour
Uterine hyper stimulation defined as more than 6 contractions by 10 minutes over a 30 minutes period | up to 2 days after cervical ripening
  uterine hyperstimulation
Requirement for tocolysis during cervical ripening or during labour | up to 2 days after cervical ripening
  requirement for tocolysis
Suspicious or pathological fetal heart rate | up to 2 days after cervical ripening
  FIGO classification
Uterine rupture | up to 2 days after cervical ripening
  yes/no
Use of analgesics during labour | up to 2 days after cervical ripening
  yes/no
Use of antibiotics during labour | up to 2 days after cervical ripening
  yes/no
Indication for caesarean delivery other than non-reassuring FHR | up to 2 days after cervical ripening
  (failure to progress in first or second stage of labour or maternal indication)
Type of vaginal delivery | up to 2 days after cervical ripening
  spontaneous or instrumental, indication for instrumental delivery
Maternal intra partum infection | up to 2 days after cervical ripening
  Suspicion of maternal intra partum infection
Maternal post partum infection | up to 2 days after cervical ripening
  Suspicion of post partum infection
Maternal post partum haemorrhage | up to 2 days after cervical ripening
  Post partum haemorrhage defined as estimated blood loss > 500 cc
Maternal blood transfusion | up to 2 days after cervical ripening
  Blood transfusion
Neonatal apgar score | at 1, 3, 5 and 10 minutes after delivery
  Apgar score at 1, 3, 5 and 10 minutes
Neonatal arterial ph | at delivery
  Arterial pH at delivery
Intensive care unit for newborn | up to 5 days after cervical ripening
  Admission in an intensive care unit
Neonatal respiratory insufficiency | up to 5 days after cervical ripening
  Respiratory insufficiency with necessity of any respiratory support
Birth asphyxia | up to 5 days after cervical ripening
  Birth asphyxia defined as pH<7, Base Excess >12 mmol/l and encephalopathy.

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - Chu Brest, Brest
  - CHU CAEN, Caen
  - Ch Pontoise, Cergy-Pontoise
  - Ch Chartres, Chartres
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Ch Departemental Vendee, La Roche-sur-Yon
  - Hopital Saint Joseph, Marseille
  - Chu Nantes, Nantes
  - Chi Poissy, Poissy
  - Chu Reims, Reims
  - Chu Rennes, Rennes
  - Chu Saint Etienne, Saint-Priest-en-Jarez
  - Chu Toulouse, Toulouse
  - Chru Tours, Tours

REFERENCES:
- [Result] Diguisto C, Le Gouge A, Arthuis C, Winer N, Parant O, Poncelet C, Chauleur C, Hannigsberg J, Ducarme G, Gallot D, Gabriel R, Desbriere R, Beucher G, Faraguet C, Isly H, Rozenberg P, Giraudeau B, Perrotin F; Groupe de Recherche en Obstetrique et Gynecologie (GROG). Cervical ripening in prolonged pregnancies by silicone double balloon catheter versus vaginal dinoprostone slow release system: The MAGPOP randomised controlled trial. PLoS Med. 2021 Feb 11;18(2):e1003448. doi: 10.1371/journal.pmed.1003448. eCollection 2021 Feb. PMID 33571294
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- [Derived] Diguisto C, Le Gouge A, Giraudeau B, Perrotin F. Mechanical cervicAl ripeninG for women with PrOlongedPregnancies (MAGPOP): protocol for a randomised controlled trial of a silicone double balloon catheter versus the Propess system for the slow release of dinoprostone for cervical ripening of prolonged pregnancies. BMJ Open. 2017 Sep 14;7(9):e016069. doi: 10.1136/bmjopen-2017-016069. PMID 28912192